CLINICAL TRIAL: NCT00001673
Title: Screening Evaluation for NIAAA Protocols
Brief Title: Screening Evaluation for Studies of the National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980009; 98-AA-0009
Record Dates: First submitted 1999-11-03; First posted 2006-04-20 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-12-15

CONDITIONS: Alcoholic Intoxication; Alcoholism; Healthy
Keywords: Alcoholics; Screening; Healthy Volunteers; Violent Abusers; Illicit Drug Testing; Blood Tests; Normal Volunteer
MeSH Terms: conditions — Alcoholic Intoxication; Alcoholism

SUMMARY:
This protocol has three purposes: (1) to evaluate subjects for inclusion or exclusion from other NIAAA protocols; (2) to provide a common set of descriptive information that will be available on all NIAAA research subjects; (3) to allow NIAAA medical and nursing staff to treat alcoholic patients for acute alcohol intoxication or alcohol withdrawal before requiring patients to consent to evaluation for participation in research studies.

Information collected will include such items as psychiatric diagnoses, presence or absence of brain, liver or other organ damage, history of the amount of past alcohol consumption, other substance use and family history of alcoholism. This information will allow investigators to determine for which, if any, NIAAA research studies a subject is eligible. In order to avoid requiring intoxicated subjects to consent for procedures such as HIV testing, psychiatric interviews, and Magnetic Resonance Imaging (MRI) of the brain we will obtain consent from all alcoholic subjects in two phases, using two separate consent forms. The first consent form will express the subject's desire to be admitted to the NIAAA inpatient unit for the purpose of treatment for alcoholism and will authorize only medical evaluation and treatment for alcoholism and associated problems. After an alcoholic subject has been admitted to the inpatient unit and is judged to be no longer intoxicated or suffering from acute alcohol withdrawal he or she will be presented with the second consent which will describe the evaluation for participation in other NIAAA research studies. Non-alcoholic, healthy controls will sign only one consent form describing the data to be collected and evaluation for participation in other NIAAA research studies.

DETAILED DESCRIPTION:
This protocol has three purposes:

1. to evaluate non-treatment seeking participants for inclusion or exclusion from other NIAAA protocols. Non-treatment seeking participants includes individuals with no current or past alcohol use disorder, as well as individuals who meet the DSM IV criteria for alcohol abuse or alcohol dependence (alcohol use disorders (AUD) but are not seeking treatment;
2. to provide a common set of descriptive information that will be available on all NIAAA research participants;
3. to collect blood samples from participants for the purpose of genetic analyses

Information collected will include such items as psychiatric diagnoses, genotypes of several neurotransmitter-related and brain growth-related candidate genes, presence or absence of brain, liver or other organ damage, history of the amount of past alcohol consumption, other substance use and family history of alcoholism. This information will allow investigators to determine for which, if any, NIAAA research studies a subject is eligible. It will also allow investigators to examine the relationship among various candidate genes and brain structure and/or function in alcoholism.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. In good health.
  2. Over 18 years of age.
  3. Not seeking treatment for alcohol or other drug use.

EXCLUSION CRITERIA:

1) Serious medical conditions that require ongoing treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2220 (Actual)
Dates: Start 1997-10-02; Study Completion 2015-12-15

CONTACTS AND LOCATIONS:
Overall Officials: Reza Momenan, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Koob GF, Nestler EJ. The neurobiology of drug addiction. J Neuropsychiatry Clin Neurosci. 1997 Summer;9(3):482-97. doi: 10.1176/jnp.9.3.482. PMID 9276849
- [Background] Heinz A, Mann K, Weinberger DR, Goldman D. Serotonergic dysfunction, negative mood states, and response to alcohol. Alcohol Clin Exp Res. 2001 Apr;25(4):487-95. PMID 11329486
- [Background] Heinz A, Ragan P, Jones DW, Hommer D, Williams W, Knable MB, Gorey JG, Doty L, Geyer C, Lee KS, Coppola R, Weinberger DR, Linnoila M. Reduced central serotonin transporters in alcoholism. Am J Psychiatry. 1998 Nov;155(11):1544-9. doi: 10.1176/ajp.155.11.1544. PMID 9812115